CLINICAL TRIAL: NCT01669005
Title: Obtaining Early Diagnosis and Prognosis in Urgent Sepsis (OEDIPUS) Study
Brief Title: The Utility of Multiplex PCR for Detection of DNA in Neutropenic Patients With Hematological Malignancies
Acronym: MedIso
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Collaborators: University Hospital, Basel, Switzerland (Other)
Responsible Party: Principal Investigator, Andrej Trampuz, MD, Centre Hospitalier Universitaire Vaudois
Other Study IDs: EK 324/06
Record Dates: First submitted 2012-08-16; First posted 2012-08-20 (Estimated); Last update posted 2012-08-20 (Estimated); Status verified 2012-08

CONDITIONS: Neutropenia
Keywords: neutropenia; multiplex PCR; infection
MeSH Terms: conditions — Neutropenia; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 3 ml of EDTA-blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Bone marrow transplant unit patients: hospitalized patients in the bone marrow transplant unit for an autologous or allogeneic hematopoietic stem cells transplantation or induction/consolidation chemotherapy

SUMMARY:
Objectives: Invasive infections are the leading cause of morbidity and mortality in patients treated for hematological malignancies. Blood cultures are often negative in neutropenic patients because of low-burden of organisms, previous antibiotic therapy or non-infectious reason of fever. More rapid, accurate and sensitive diagnostic tools are needed.

Hypothesis: Multiplex real-time PCR may detect microbial DNA in neutropenic patients before febrile episode. To investigate this hypothesis, EDTA-blood was routinely collected for multiplex PCR at admission and 3x/week thereafter until discharge or recovery from neutropenia

ELIGIBILITY:
Inclusion Criteria:

* patients aged ≥18 years
* autologous or allogeneic hematopoietic stem cells transplantation or induction/consolidation chemotherapy performed

Exclusion Criteria:

* No blood samples were taken

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients hospitalized in the bone marrow transplant unit in the study period
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2007-11; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrej Trampuz, MD, Study Director — University Hospital Lausanne, Switzerland; Christina Orasch, MD, Principal Investigator — University Hospital Lausanne, Switzerland